CLINICAL TRIAL: NCT06014996
Title: Pulsed Field Ablation Using a Novel Biphasic Catheter vs Thermal Ablation for Paroxysmal Atrial Fibrilation:InsightPFA Trial
Brief Title: InsightPFA Trial of the LotosPFA Catheter
Acronym: InsightPFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insight Medtech Co., Ltd. (Industry)
Collaborators: Insight Lifetech Co., Ltd. (Industry); Guangdong Provincial People's Hospital (Other); Beijing Anzhen Hospital (Other); Sir Run Run Shaw Hospital (Other); Shanghai Zhongshan Hospital (Other); The Affiliated People's Hospital of Ningbo University (Other Government); The First Affiliated Hospital of Dalian Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Weifang People's Hospital (Other)
Responsible Party: Sponsor
Organization: Insight Lifetech Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101000001M-CIP-001
Record Dates: First submitted 2023-08-07; First posted 2023-08-28 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Arrhythmias, Cardiac; Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; pulmonary vein isolation; pulsed field ablation; randomized controlled trial
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: symptomatic paroxysmal AF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Test group will utilize the cardiac PFA system (including a pulsed field generator, an expandable PFA catheter, and a steerable sheath) from Insight Medtech.
  Interventions: Device: Pulsed Field Ablation (PFA) Therapy
- Control group (Active Comparator): The control group will utilize an RFA system (including CARTO VISITAG Module and the THERMOCOOL SMARTTOUCH Catheter) from Biosense Webster.
  Interventions: Device: Radiofrequency Ablation（RAF）Therapy

INTERVENTIONS:
Device: Pulsed Field Ablation (PFA) Therapy — In the test group, subjects will undertake PVI using the PFA system including a nanosecond-scale pulsed field generator (InRythm, Insight Lifetech, Shenzhen, China), a lotos catheter that is expandable over the wire (LotosPFA, Insight Lifetech), and a customized 12-French steerable sheath (InBridge, Insight Lifetech).
  Arms: Test group
Device: Radiofrequency Ablation（RAF）Therapy — In the control group, subjects will undergo PVI using an RFA system including CARTO VISITAG Module and the THERMOCOOL SMARTTOUCH Catheter (Biosense Webster Inc., Diamond Bar, CA, USA). PVI was performed with AI values of 400-450 in the anterior, 300-350 at the posterior wall of the LA.
  Arms: Control group

SUMMARY:
This trial aims to determine whether the InsightPFA for PVI is as effective and safe as standard RFA in the treatment of symptomatic paroxysmal AF.

DETAILED DESCRIPTION:
The InsightPFA trial is a prospective, multicenter, randomized controlled trial to compare the effectiveness and safety of PFA versus RFA for PVI in Chinese patients with symptomatic paroxysmal AF. Two hundred and ninety-two patients diagnosed with symptomatic paroxysmal AF will be randomly assigned to either the PFA group or the RFA group in a 1:1 ratio. All subjects will undergo PVI using PFA or AI guided RFA and be followed up to 12 months. The primary endpoint is defined as freedom from any episodes of AF/AFL/AT without Class I or III antiarrhythmic drugs during the 9-month follow-up period after a 90-day blank period. The secondary endpoints of effectiveness include acute treatment success and procedural data. The safety evaluation includes a composite of death, stroke and transient ischemic attack, procedure-related complications, device-related adverse events, and serious adverse events. A noninferiority comparison will be conducted between the novel PFA system and the existing RFA system in terms of both effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, of either sex.
2. Patients with ECG-confirmed or clinically definite diagnosis of symptomatic paroxysmal atrial fibrillation (PAF).
3. Scheduled to undergo catheter ablation for atrial fibrillation
4. Willing to participate in this clinical trial, voluntarily sign the informed consent form, and commit to completing required examinations and follow-ups per protocol..

Exclusion Criteria:

1. History of prior surgery or catheter ablation for atrial fibrillation (AF);
2. Clinical diagnosis of persistent or long-standing persistent AF;
3. Left ventricular ejection fraction (LVEF) < 40% or New York Heart Association (NYHA) functional class III or IV;
4. Left atrial diameter (as measured by echocardiography) ≥ 50 mm;
5. Imaging findings suggestive of left atrial or left atrial appendage thrombus;
6. Contraindications to anticoagulation therapy, including a history of blood clotting disorders or abnormal bleeding;
7. Presence of acute or active systemic infection;
8. Significant lung disease, pulmonary hypertension, or any lung condition associated with severe dyspnea, such as abnormal blood gases;
9. Clinical diagnosis of hypertrophic cardiomyopatly, chronic obstructive pulmonary disease (COPD), or known/suspected atrial myxoma;
10. History of previous heart valve repair or replacement, implantation of a prosthetic valve, or previous cardiac interventions such as atrial septal defect closure or patent foramen ovale closure;
11. Presence of an implanted cardioverter defibrillator or other active implanted devices;
12. Myocardial infarction, unstable angina, or any cardiac intervention/open surgery (excluding coronary angiography) within the past 3 months; hospitalization for heart failure, stroke (excluding silent stroke), or transient ischemic attack within the past 3 months;
13. Any carotid stenting or endarterectomy performed within the past 6 months;
14. Patients who have clear contraindications to interventional procedures, rendering them unsuitable for the ablation procedure in the judgment of the investigator;
15. Participation in other drug or device clinical trials concurrently;
16. Life expectancy of less than 12 months due to conditions such as advanced malignancy;
17. Women who are pregnant, breastfeeding, or planning to conceive during the trial period;
18. Any other situations deemed inappropriate for participation in the clinical trial as determined by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
the 12-month treatment success rate | during the 12-month follow-up period after a 90-day blank period.
  12month treatment success, is defined as freedom from any episodes of AF/atrial flutter (AFL)/atrial tachycardia (AT) without the use of Class I or III antiarrhythmic drugs (AADs) during the 12-month follow-up period after a 90-day blank period. An electrocardiogram or 24 h Holter monitoring should be performed to confirm all episodes.
  The occurrence of AF/AFL/AT during a blank period is not considered a treatment failure and can be treated with AADs (other than amiodarone), electric cardioversion, or only a time of catheter ablation procedure (the devices used during the redo procedure should be the same as those used in the original procedure). After the blanking period, any documentation of AF, AFL, or AT ≥ 30 s is considered a failure concerning the primary effectiveness endpoint. Following the blanking period, any use of a Class I or III AAD constitutes a treatment failure.

SECONDARY OUTCOMES:
Acute procedural success | after a 20 min observation period following the last ablation.
  Acute procedural success is defined as the isolation of each PV after a 20 min observation period following the last ablation.
Total procedure time | During the procedure
  Procedure duration in minute
Total left atrium indwelling time | During the procedure
  Procedure duration in minute
Total abaltion time | During the procedure
  Procedure duration in minute
Total X-ray exposure time | During the procedure
  Total time of X-ray exposure
Total X-ray exposure dose | During the procedure
  Total dose of X-ray exposure
Number of participants under general anesthesia | During the procedure
  Comparison of number of patients under general anesthesia between two groups.
Evaluation of the ablation system（questionnaire） | immediately post ablation
  To evaluate the stability of both systems concluded from all enrolled case using questionnaire, including below measures :
  1. the stability of the ablation system ;
  2. the usability of the ablation system .
  For each system in 1., 2., and 3., only one of the following five ratings is given:
  1. very stable;
  2. stable, inspection was unaffected;
  3. slightly unstable, inspection was unaffected;
  4. N/A.
Evaluation of the ablation catheter（questionnaire） | immediately post ablation
  To evaluate the maneuvering performance of catheters in the two systems concluded from all enrolled case, including below measures :
  1. whether the ablation catheter can reach the expected position smoothly for ablation；
  2. whether the ablation catheter can be visible clearly under X-ray；
  3. whether the energy of the ablation catheter cannot be released after system operation
Evaluation of the adjustable introducer sheath set（questionnaire） | immediately post ablation
  To evaluate the adjustable introducer sheath set of the investigation device， including below measures :
  1. whether the introducer sheath can reach the expected position smoothly for ablation；
  2. whether the introducer sheath can be visible clearly under X-ray；
  3. whether the curved shape of the introducer sheath can be adjustable。
incidence of composite safety endpoint | 12 months after the ablation
  Composite safety endpoint composed of: procedure-related deaths, strokes, and transient ischemic attacks
incidence of surgical complications | 12 months after the ablation
  surgical complications composed of: vascular puncture/bleeding complications, cardiac tamponades and/or perforations, left atrial-esophageal fistula, phrenic nerve injury, and pulmonary vein stenosis
Incidence of severe adverse events | 12 months after the ablation
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.
Incidence of device-related adverse events | 12 months after the ablation
  Device-related adverse events refer to an adverse medical event related to the use of a device that occurs during the course of the clinical trial. However, a distinction should be made with respect to normal postoperative stress response, such as fever and chest and back discomfort, which, in the judgment of the investigator, need not be recorded as an adverse event. Recording of device-related adverse events will be applicable for conditions that are deemed by the investigator to be definitely related, possibly related, or of indeterminate relationship, to the test device.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital, Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Yan'an Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Hanzhou, Zhejiang
  - The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin W, Chu H, Wang C, Chang D, Yin X, Wang Y, Jiang C, Xu Y, Liao Q, Yang J, Zhu W, Li S, Gao W, Chen Y, Yu Y, Li Q, Liao H, Deng H, Wei W, Pu S, Guo Z, Xu D, Li W, Ouyang F, Xue Y; InsightPFA Investigators. Pulsed Field Ablation Using a Novel Biphasic Catheter vs Thermal Ablation for Paroxysmal Atrial Fibrillation: InsightPFA Trial. J Am Coll Cardiol. 2025 Dec 9;86(23):2314-2326. doi: 10.1016/j.jacc.2025.09.1593. PMID 41338842
- [Derived] Lin W, Pu S, Chu H, Chang D, Yin X, Wang Y, Xu Y, Li S, Yang J, Zhu W, Li S, Gao W, Chen Y, Xu D, Jiang C, Xue Y. Rationale and Design of the InsightPFA Trial: A Prospective, Multicenter, Randomized Controlled Trial of the Irreversible Electroporation-Based Pulsed Field Ablation Versus Radiofrequency Ablation in Chinese Patients With Symptomatic Paroxysmal Atrial Fibrillation. J Cardiovasc Electrophysiol. 2025 Mar;36(3):632-641. doi: 10.1111/jce.16573. Epub 2025 Jan 24. PMID 39853845